CLINICAL TRIAL: NCT05696769
Title: Measuring Stigmatization in Chronic Tic Disorders: Development and Validation of the Tourette Discrimination-Stigmatization (TD-STIGMA) Scale
Brief Title: Tourette Discrimination (TD) Stigma Scale
Acronym: TD
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Tourette Association of America (Other); University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00080472
Record Dates: First submitted 2023-01-12; First posted 2023-01-25 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Tourette Syndrome; Tourette Syndrome in Children; Tourette Syndrome in Adolescence; Tic Disorder, Childhood; Tics
Keywords: Stigma
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders; Tics; Social Stigma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Youth with CTD Ages 8-12: Youth (8-12 years) will be recruited for a qualitative interview using the exploratory questionnaire developed for the study. Parent/caregivers will also be asked questions related to their child's CTD. Participants will be asked for feedback on the ease of completion, content, readability and completion time.
  After development of the TD Stigma scale, prior and new participants with CTD will be asked to complete the TD-Stigma scale with companion measures. Feedback on the scale will be elicited as well.
- Supporters: Parents/Caregivers: Qualitative interviews will be administered and adapted to the caregiver's perspective. Parents/caregivers will also be asked to complete questionnaires child's CTD history, family history and impact of CTD on different aspects of the child's life. Participants will be asked for feedback on the ease of completion, content, readability and completion time.
- Provider/ advocate cohort: For providers and advocates, qualitative interview administered will begin with the participant's experience and qualifications in caring for individuals with CTD and adapted to the provider's perspective. Participants will be asked for feedback on the ease of completion, content, readability and completion time.
- Youth with CTD Ages 13-17: Youth (13-17 years) will be recruited for a qualitative interview using the exploratory questionnaire developed for the study. Parent/caregivers will also be asked questions related to their child's CTD. Participants will be asked for feedback on the ease of completion, content, readability and completion time.
  After development of the TD Stigma scale, prior and new participants with CTD will be asked to complete the TD-Stigma scale with companion measures. Feedback on the scale will be elicited as well.
- Adults with CTD Ages (18-30): Adults with CTD (Ages 18-30) will be recruited for a qualitative interview using the exploratory questionnaire developed for the study.
  Participants will be asked for feedback on the ease of completion, content, readability and completion time.
  After development of the TD Stigma scale, prior and new participants with CTD will be asked to complete the TD-Stigma scale with companion measures. Feedback on the scale will be elicited as well.
- Supporters: Partners/Spouses/Significant others: For Partners/Spouses/Significant others, qualitative interview administered will begin with the participant's experience and qualifications in caring for individuals with CTD and adapted to the supporter's perspective. Participants will be asked for feedback on the ease of completion, content, readability and completion time.

SUMMARY:
The goal of this qualitative study is to understand the challenges of stigmatization and discrimination in children and young adults with Chronic Tic Disorders (CTD), including Tourette Syndrome. Measuring and understanding how stigma affects those with CTD will help inform future work.

DETAILED DESCRIPTION:
This study will utilize a phased approach, where (1) Narrative and thematic content data will be obtained through in-depth qualitative interviews of CTD stakeholders. (2) Based on these results, a novel scale will be developed through the Delphi Method with CTD stakeholders. (3) Preliminary analyses of the scale's psychometric properties.

ELIGIBILITY:
Inclusion Criteria:

CTD Cohort

1. Physician-confirmed diagnosis of CTD based on the Diagnostic and Statistical Manual for Mental Disorders-Fifth Edition (DSM-V) criteria
2. 8-30 years old.

Parent/caregivers, supporters, medical providers, advocate cohort (s)

1. Involved in the care of a child, youth or young adult with CTD
2. The known person with CTD has had tics for more than a year at the time of screening

Exclusion Criteria:

CTD Cohort

Exclusion criteria:

1. Non-English speaking
2. Diagnosis of intellectual disability
3. Diagnosis of psychosis
4. Any other condition that, in the Principle Investigator's opinion, would limit the participant's (or parent's) ability to understand study measures.

Parent/caregivers, supporters, medical providers, advocate cohort (s)

1) The known person with CTD has an intellectual disability or diagnosis of psychosis

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Youth and Young adults with CTD (Chronic Tic Disorder, Tourette) Supporters of individuals with CTD - parents or caregivers, partners Providers/advocates of individuals with CTD - clinicians, therapists, patient advocacy group representatives
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2023-03-04 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Change in Tourette Discrimination-Stigmatization (TD-STIGMA) scores | Month 7
  Confirmatory factor analysis will be used to assess the factor structure of the hypothesized domains. Mean TD-STIGMA scores will be calculated. Internal consistency (both overall and within each domain) will be evaluated using Cronbach's alpha. Intraclass correlation will be used to evaluate test-retest reliability by retesting a subset of participants (n=20) two weeks after test administration. Some items may be removed from the list based on the results of the factor analysis, internal consistency, and test-retest evaluation. Both convergent validity and known-group validity will be evaluated. Analyses will use SAS 9.3.

OTHER OUTCOMES:
Qualitative Interviews | 3 hours
  Stakeholder interviews will be audio-recorded, transcribed, and input into NVivo software for qualitative analysis. Transcripts will be compared with original recordings to ensure accuracy. Interviews will be analyzed using deductive thematic content analysis practices to identify emerging themes and subthemes.
Tourette Discrimination-Stigmatization (TD-STIGMA) Scale psychometric properties | Month 4
  A de-identified summary document of thematic content and narrative content analysis from Aim 1 will be securely emailed to stakeholders. Content will be alphabetized to avoid introducing bias. Stakeholders will be blind-copied to maintain anonymity. Using the Delphi Method, they will be asked to prioritize responses, provide feedback and propose solutions. The feedback process will continue until there is an 80% consensus among stakeholders. The outcome will be a close-ended TD-STIGMA scale. The Flesch Reading Ease score and Flesch-Kincaid Grade level will be used to assess questionnaire readability.

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn M Martindale, DO, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentified
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent re view committee ("learned intermediary") identified for this purpose. For individual participant data meta-analysis. Proposals should be directed to the study PI jmartind@wakehealth.edu

REFERENCES:
- [Derived] Martindale JM, Chapman L, Carson AJ, Reilly K, Malli M, Storch EA, Salsman J, Daniel S. Beyond the Tics: Experiences of Stigma and Psychosocial Impact in Tourette Syndrome. Child Psychiatry Hum Dev. 2026 Jan 24. doi: 10.1007/s10578-026-01965-0. Online ahead of print. PMID 41579326